CLINICAL TRIAL: NCT04391335
Title: Novel Pulmonary Function Measures for Diagnosis of Bronchiolitis Obliterans Syndrome Following Hematopoietic Stem-Cell Transplantation in Children
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Giles Santyr, Senior Scientist, The Hospital for Sick Children
Other Study IDs: 1000063459
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Bronchiolitis Obliterans Syndrome
Keywords: Stem cell transplantation; Xenon MRI; Lung
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Participants who meet the screening criteria for the development of bronchiolitis obliterans syndrome (BOS) according to the NIH criteria
- Group 2: Participants who may or may not have abnormal spirometry; however they do not fulfill the NIH criteria for the development of BOS

SUMMARY:
In this study, we will study 129Xe-MRI and LCI as tools for diagnosis of BOS in pediatric patients who have received Hematopoietic Stem Cell Transplantation (HSCT) and have been identified as eligible for this study. Participants will be required to have vital signs collected, complete breathing tests and complete an MRI. The MRI will require participants to perform breath holds in the MRI scanner with xenon gas while being coached by a research assistant.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 6 -17.9 years old.
* Received HSCT treatment at least 6 months prior to enrollment in study.
* Participants should have an FEV1%pred value greater than 40%.
* Participant understands the study procedures and is willing to participate in the study as indicated by signature on the informed consent or assent.
* Participant must be able to perform a breath hold for 16s.
* Participant meets MRI screening criteria

Exclusion Criteria:

* Participant has had a cold or respiratory infection in the last four weeks.
* Participant requires supplemental oxygen or has a daytime room air oxygen saturation ≤ 95%.
* Participant is unable to perform spirometry or plethysmography maneuvers.
* Participant is pregnant or lactating.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Two groups of participants will be recruited. Group 1 will be participants who meet the screening criteria for the development of BOS according to the NIH criteria. Group 2 will be participants who may or may not have abnormal spirometry; however they do not fulfill the NIH criteria for the development of BOS.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of MRI | 24 months
  Perform xenon MRI, in participants with and without a diagnosis of BOS as defined by NIH criteria.

SECONDARY OUTCOMES:
Correlation | 24 months
  Correlate MRI with conventional breathing tests

CONTACTS AND LOCATIONS:
Overall Officials: Giles Santyr, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No